CLINICAL TRIAL: NCT02533141
Title: Effect of Simvastatin Withdrawal on Ocular Endothelial Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-240215
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Investigation of the changes of flicker induced vasodilatation before, during and after withdrawal of therapy with simvastatin
MeSH Terms: interventions — Laser-Doppler Flowmetry; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 10 healthy subjects receiving at first simvastatin for 4 weeks, then crossover. Measurements will be done with the Dynamic Vessel Analyzer (DVA) and Laser Doppler Velocimetry (LDV).
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Laser Doppler Velocimetry (LDV); Drug: Simvastatin
- Placebo group (Placebo Comparator): 10 healthy subjects receiving at first placebo for 4 weeks, then crossover. Measurements will be done with the Dynamic Vessel Analyzer (DVA) and Laser Doppler Velocimetry (LDV).
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Laser Doppler Velocimetry (LDV); Other: Placebo

INTERVENTIONS:
Device: Dynamic Vessel Analyzer (DVA) — Measurement of flicker induced vasodilatation, retinal vessel diameters and oxygen saturation
Device: Laser Doppler Velocimetry (LDV) — Measurement of red blood cell velocity in retinal vessels
Drug: Simvastatin — Simvastatin Ranbaxy (Basics GmbH, Leverkusen, Germany) Dosage: 40 mg per day for 4 weeks, ingested in the morning Route of administration: peroral
  Arms: Intervention group
Other: Placebo — Placebo, once daily for 4 weeks
  Arms: Placebo group

SUMMARY:
Statins are drugs representing the most commonly prescribed medication for the treatment of hypercholesterolemia. In a recently published study, discontinuation of statin therapy in patients after acute myocardial infarction was associated with a higher all-cause mortality (hazard ratio 3,45) and a higher cardiac mortality (hazard ratio 4,65). Increasing evidence suggests that statins also have vasoactive properties by up-regulating endothelial nitric oxide synthase (eNOS) with positive effects on endothelial function. Experiments with flow-mediated vasodilatation (FMD) showed these positive effects of statin treatment on endothelial function but also revealed that withdrawal of statin treatment transiently worsens endothelial function, independently of serum cholesterol levels.

Consequently, this placebo controlled Phase IV crossover study wants to assess changes of endothelial function in terms of flicker induced vasodilatation before and during statin therapy as well as after statin withdrawal. For this purpose 20 healthy subjects will be treated with 40 mg/day of simvastatin for a period of 4 weeks. Flicker induced vasodilatation and retinal oxygen saturation will be measured with the Dynamic Vessel Analyzer system by Imedos at baseline, in the 4th week of simvastatin or placebo intake as well as 3, 7 and 14 days after the end of intake.

ELIGIBILITY:
Inclusion Criteria:

Informed consent for participation

* Men and women aged between 18 and 45 years, non-smokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg
* Normal ophthalmic findings, ametropia less than 6 diopters

Exclusion Criteria:

* History or presence of ocular disease
* Ametropy ≥ 6 dpt
* Previous or current treatment with statins
* Treatment with any drug in the 3 weeks preceding the first study day
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Participation in a clinical trial in the 3 weeks preceding the first study day
* Blood donation during the 3 weeks preceding the first study day
* History or family history of epilepsy
* History or presence of myopathy, renal failure or elevation of creatine kinase (CK) above normal levels
* History or presence of hepatic dysfunction, including increase of liver enzymes
* Abuse of alcoholic beverages
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Flicker induced vasodilatation (DVA) | 16 weeks

SECONDARY OUTCOMES:
Retinal oxygen saturation (DVA) | 16 weeks
Red blood cell velocity (LDV) | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria